CLINICAL TRIAL: NCT04624620
Title: A Culinary-Based Intensive Lifestyle Program for Patients With Obesity
Acronym: TKCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Auden McClure, Assistant Professor in Pediatrics, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20143
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot (Experimental): Participants will participate in a 16 week, culinary intensive study that will consist of 2 hour virtual classes taught by a chef, a dietitian, and a health coach that focus on diet, culinary competency, daily physical activity, mindfulness and support for behavior change.
  Interventions: Behavioral: Teaching Kitchen Collaborative Curriculum

INTERVENTIONS:
Behavioral: Teaching Kitchen Collaborative Curriculum — This is a referral-based teaching kitchen intervention that synergistically provides basic cooking skills, an evidence-based nutrition curriculum, mindfulness skills, activity tracking, and support for behavior change to augment weight management and lifestyle change in the primary care setting.

SUMMARY:
The study team proposes in this pilot to test, in a single-arm mixed-methods study, the feasibility, acceptability, and preliminary effectiveness of the 16 modular classes taught by a chef, dietitian, and health coach. While the pilot may not have the power to detect significant change, it will provide preliminary data for a NIH application to further test this curriculum in a pragmatic, community-based, randomized multi-site Teaching Kitchen Collaborative Curriculum (TKCC) study planned for Jan 2022 or thereafter. If effective, the TKCC has potential to impact population health through translation into teaching kitchens nationally and adaptation to clinic /community settings.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* English speaking patients
* Aged 30-65 (in order to capture adults living independently)
* Diagnosis of class I or II obesity (BMI 30-39.9 kg/m2)
* Participants must be available for and willing to commit to the sixteen classes either in person or virtually.
* Must have a device with a camera (smartphone, tablet, computer)
* Use email and text
* Home Wi-Fi with high-speed internet
* Must have minimal cooktop and oven capacity at home
* Participants will be referred AND have medical clearance from a primary care provider at Dartmouth-Hitchcock

Exclusion Criteria:

* Patients taking obesity or diabetes medications as assessed by study medical director
* severe obesity (BMI≥40kg/m2)
* Diagnosis of Type 2 diabetes (HA1C ≥ 6.5) in the past (excluding gestational diabetes)
* implanted electronic medical device
* History of bariatric surgery
* Current participation in a longitudinal culinary or weight management program, including the D-H Weight and Wellness Center
* Severe mental health or life-threatening illnesses
* Unstable cardiovascular disease
* Hospitalization for depression in past 6 month
* Self-report of alcohol or substance abuse within the past 12 months
* Diet / exercise contraindications
* Other medical, psychiatric, or behavioral limitations that in the judgment of the principal investigator may interfere with study participation or the ability to follow the intervention protocols determined by PI
* Prisoners
* Pregnant women will not be eligible to participate nor will those unable or unwilling to give informed consent or communicate with local study staff.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Program Feasibility based on program attendance | 16 weeks
  Number of classes Participants attend
Program Feasibility based on Completion rate | 16 weeks
  Calculated using the following formula: (# completing all classes / # enrolled).
Program Feasibility based on Assessment Completion rate | 16 Weeks
  Calculated using the following formula: (# completing all assessments / # enrolled).
Program Feasibility based on Enrollment rate | 16 weeks
  Calculated using the following formula: [# enrolled / (# referred & eligible)].
Program Feasibility based on Number of withdrawals (dropouts) | 16 Weeks
  Number of enrolled participants officially withdrawing from the study and reason for withdrawal
Program Feasibility based on Number lost to follow up (attrition) | 16 Weeks
  Number who failed to attend sessions and could not be contacted for follow-up
Program Acceptability based on participant interviews evaluating the pilot and assessing strengths/weaknesses. | 16 weeks
  Program acceptability will be assessed through participant semi-structured participant interviews assessing program strengths/weaknesses.
Program Acceptability based on participant surveys | 16 weeks
  Program acceptability will be assessed through participant surveys assessing program strengths/weaknesses. Based on [1-5] likert scale.

SECONDARY OUTCOMES:
Change in Body Weight | Baseline, 16 weeks, 1 year
  kg
Change in Body Mass Index | Baseline, 16 weeks, 1 year
  Height (cm) and Weight (kg) will be used to calculate body mass index (kg/m^2)
Change in Waist Circumference | Baseline, 16 weeks
  Waist circumference will be measured (cm)
Change in Percent Body Fat | Baseline, 16 weeks
  Percent Body Fat
Change in Visceral fat area | Baseline, 16 weeks
  Visceral fat area (cm2)
Change in skeletal muscle mass | Baseline, 16 weeks
  skeletal muscle mass (lbs)
Change in TKCC Survey Responses | Baseline, 16 Weeks
  The Teaching Kitchen Collaborative Curriculum (TKCC) survey is an investigator created, non-validated Health Habits Survey that assesses nutrition, exercise, cooking habits, sleep behaviors, basic medical information, readiness to change, mindfulness, and telehealth experience. Individual survey questions have variable response categories (examples: commitment to change) is assessed using a 1 to 10 scale with 1 being a less favorable response, and 10 is a more favorable response.
Change in Mindfulness | Baseline, 16 Weeks
  The Mindful Easting Questionnaire (MEQ) is a widely used instrument that assesses trait mindfulness.
Change in Quality of Life | Baseline, 16 Weeks
  Short Form RAND Survey. Quality of life will be assessed using the 20-item Short Form Survey Instrument (SF-20). It was developed by the RAND corporation. The SF-20 is a well accepted and valid survey used to assess overall health measuring 8 different dimensions including physical and social functionality and limitations, mental health, vitality, pain, general health perception, and health change.
Change in Readiness to Change | Baseline, 16 Weeks
  University Rhode Island Change Assessment Scale (URICA). Self-reported survey of respondents' feelings about changing their weight problem. Total score is also called the Readiness Score, ranging from -2 to +14 (worse to better), calculated by subtracting the mean from the precontemplation responses from the summation of the means of responses to contemplation, action, and the struggling to maintain items.
Change in Nutrition | Baseline, 16 Weeks
  US PDQS. As measured by participants self-reported eating habits on fruits, vegetables, and other diet habits.Scores associated with the healthier dietary pattern are higher and lower for unhealthy patterns.
Change in Food Insecurity | Baseline, 16 Weeks
  Hunger Vital Signs. 2-questions to assess food insecurity as recommended by the American Academy of Pediatrics:
  "We worried whether our food would run out before we got money to buy more." Was that often true, sometimes true, or never true for your household in the last 12 months? "The food we bought just didn't last, and we didn't have money to get more." Was that often true, sometimes true, or never true for your household in the last 12 months? A response of "often true" or "sometimes true" to either question = positive screen for Food Insecurity.
Self Efficacy for Eating/Cooking Fruit and Vegetables by Condrasky | Baseline, 16 Weeks
  Cooking attitudes as measured by self reported attitudes about cooking and the use of the provided fresh fruits and vegetables to provide food to themselves and or their families.
Change in Sleep | Baseline, 16 Weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep
Change in Exercise | Baseline, 16 Weeks
  Exercise vital sign: (EVS is calculated by multiplying responses to "On average, how many days per week do you engage in moderate to strenuous exercise (like a brisk walk)?" and 2) "On average, how many minutes per day do you engage in exercise at this level?" in order to display minutes per day of moderate or strenuous exercise.
Change in Fasting glucose | Baseline, 16 weeks
  Fasting glucose mg/dl
Change in Fasting Insulin | Baseline, 16 weeks
  Fasting insulin mg/dl
Change in Fasting Lipid Profile | Baseline, 16 weeks
  Cholesterol mg/dl
Change in Hemoglobin A1c | Baseline, 16 weeks
  Hemoglobin A1c mmol/mol
Change in ALT | Baseline, 16 weeks
  Hemoglobin ALT mg/dl
Change in AST | Baseline, 16 weeks
  Hemoglobin AST mg/dl
Change in Microbiome | Baseline, 16 weeks
  stool samples

OTHER OUTCOMES:
Staff Adoption | 16 weeks
  Qualitative semi-structured interviews will ensure the appropriateness of the pilot and its strengths/weaknesses.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No